CLINICAL TRIAL: NCT07164157
Title: The Risk of Adverse Pregnancy Outcomes for Long-term Exposure to Air Pollution in Pregnant Patients With Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Wei Huang (Other)
Responsible Party: Sponsor-Investigator, Wei Huang, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025XMSB0000311
Record Dates: First submitted 2025-03-12; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Arterial Hypertension; Air Pollution; Maternal Outcome
Keywords: pulmonary hypertension; air pollution; maternal outcome; heart failure; preterm birth; low birth weight
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Heart Failure; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (24):
- The First Affiliated Hospital of Chongqing Medical University
- The Second Affiliated Hospital of Chongqing Medical University
- Xiangya Hospital of Central South University
- The second Xiangya Hospital of Central South University
- Yan'an Hospital of Kunming City
- Gansu Provincial Hospital
- Qilu Hospital of Shandong University
- The second hospital of Army Military University
- Guizhou Provincial People's Hospital
- The Second Affiliated Hospital of Nanchang University
- Henan Provincial People's Hospital
- Gannan Medical University
- Women and Children's Hospital of Chongqing Medical University
- The First People's Hosipital of Yunnan Province
- People's Hosipital of Xinjiang Uygur Autonomous Region
- The First Affiliated Hospital of Anhui Medical University
- Yantai Yuhuangding Hospital
- The Third People's Hosipital of Chengdu
- Zhongda Hospital Southeast University
- The First Affiliated Hospital of Xi'an Jiao Tong University
- Gansu Provincial Maternity and Child-care Hospital
- The First Affiliated Hospital of Guangxi Medical University
- Xijing Hospital
- Shenzhen People's Hospital

SUMMARY:
With economic development and rapid urbanization, air pollution has become an increasingly severe public health concern. The risk of adverse pregnancy outcomes is significantly elevated for pregnant women complicated by pulmonary hypertension. However, no studies to date have specifically examined the impact of environmental factors on pulmonary hypertension in pregnant women, nor their subsequent birth outcomes. Therefore, investigating the correlation between them holds substantial clinical and public health significance.

DETAILED DESCRIPTION:
The purpose of the research is preliminary found that the correlation between air pollution and maternal outcomes in pregnant women with pulmonary arterial hypertension and provide useful information for managment of pregnant women in special ambient conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with pulmonary hypertension who attended major medical centers included in this study from January 2013 to December 2022.

  * Complete medical records available; ② Pulmonary artery systolic pressure ≥ 35 mmHg by echocardiography or a confirmed diagnosis of pulmonary hypertension by right heart catheterization; ③ Residential address information available at the city (district, county) level or higher.

Exclusion Criteria:

* ① Unclear diagnosis and completely missing address information;

  * Incomplete medical records; ③ Lost to follow-up during pregnancy or within six weeks postpartum.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with pulmonary hypertension(PH) who attended major medical centers included in this study from January 2013 to December 2022. Our study includes all types of pregnant women with PH, primarily those who with congenital heart disease-associated PH, followed by those with left heart disease-associated PH.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
1.main maternal outcome | diagnosis of pregnancy to six months postpartum
  including maternal death and heart failure

SECONDARY OUTCOMES:
Secondary maternal outcome events | From delivery to 42 days postpartum
  including other cardiac events: arrhythmia requiring treatment, thromboembolic event, myocardial infarction, stroke, pulmonary hypertension crisis and so on.

OTHER OUTCOMES:
2.main offspring events | From delivery to 42 days postpartum
  including fetal or neonatal death, prematurity, low birth weight, small for gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided